CLINICAL TRIAL: NCT01333605
Title: Phase II Study of IGEV Followed by Autologous Stem Cell Transplantation in Patients With Refractory or Relapsed Hodgkin Lymphoma.
Brief Title: IGEV Followed by Autologous Transplantation for Refractory or Relapsed Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 11-02
Record Dates: First submitted 2011-04-11; First posted 2011-04-12 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2013-03

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin lymphoma; Chemotherapy; IGEV; Autologous stem cell transplantation
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IGEV regimen (Experimental): Ifosfamide 1200 mg/m2 at days 1-4, Mesna 400 mg 0,4,8h at days 1-4, Gemcitabine 800 mg/m2 at day 1 and day 4, Vinorelbine 20 mg/m2 at day 1, Prednisone 100 mg at days 1-4. Frequency of cycles: every 3 weeks. Numbers of cycles: 4 cycles
  Interventions: Drug: IGEV

INTERVENTIONS:
Drug: IGEV — Ifosfamide 1200 mg/m2 at days 1-4, Mesna 400 mg 0,4,8h at days 1-4, Gemcitabine 800 mg/m2 at day 1 and day 4, Vinorelbine 20 mg/m2 at day 1, Prednisone 100 mg at days 1-4. Frequency of cycles: every 3 weeks. Numbers of cycles: 4 cycles.

SUMMARY:
The aim of study is to prove IGEV regimen followed by autologous stem cell transplantation as salvage treatment in patients with refractory or relapsed Hodgkin lymphoma is effective.

DETAILED DESCRIPTION:
The standard treatment in patients with refractory or relapsed Hodgkin lymphoma is salvage chemotherapy followed by autologous transplantation for responsive patients. However, the standard of salvage chemotherapy remains uncertain. This study is to evaluate the efficacy and safety of IGEV regimen in a single-center basis.

ELIGIBILITY:
Inclusion Criteria:

* Age range: 18-65 years old
* Histological confirmed refractory or relapsed Hodgkin lymphoma
* With at least one site of measurable disease according to IWC criteria
* ECOG performance status 0-1
* Life expectancy of more than 3 months
* Bone marrow function: ANC≧1.5×109/L, PLT≧100×109/L, Hb≧80g/L
* Liver function: total bilirubin, ALT and AST <1.5×UNL
* Renal function: Cr<1.5×UNL, CCR≧45ml/min
* No contraindication for transplantation

Exclusion Criteria:

* No prior chemotherapy
* With more than 2 lines of prior chemotherapy exposure
* Evidence of CNS and bone marrow involvement
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Significant active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2011-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 6 weeks

SECONDARY OUTCOMES:
Overall response rate | 6 weeks
3-year progression-free survival rate | 3 years
3-year overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China